CLINICAL TRIAL: NCT00325143
Title: Assess Safety & Reactogenicity of DTPa-IPV/Hib Vaccine Admnd at 3 & 4 Mths & DTPa-HBV-IPV/Hib Vaccine Admnd at 5 Mths, Followed by DTPa-IPV/Hib Vaccine at 18 Mths in Infants Who Received hepatitisB Vaccine at Birth & at One Month of Age
Brief Title: Safety of DTPa-IPV/Hib & DTPa-HBV-IPV/Hib, Followed by DTPa-IPV/Hib Vaccine in Infants Who Received Hepatitis B Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 217744/100
Record Dates: First submitted 2006-02-08; First posted 2006-05-12 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Haemophilus Influenzae Type b; Diphtheria; Tetanus; Poliomyelitis; Acellular Pertussis
MeSH Terms: conditions — Haemophilus Infections; Diphtheria; Tetanus; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (1):
- Infanrix Hexa Group (Experimental): Healthy male or female subjects between and including 11 to 17 weeks of age, who were previously vaccinated with Rotarix™ in study 444563/028 (NCT00197210), additionally received 2 doses of Infanrix™-IPV/Hib vaccine (at 3 and 4 months of age), 2 doses of Rotarix™ vaccine (at 2 and 4 months of age) and one dose of Infanrix Hexa™ vaccine (at 5 months of age) as a primary vaccination course, followed by administration of a booster dose of Infanrix™-IPV/Hib vaccine (at 18 months of age). The Infanrix™-IPV/Hib and Infanrix Hexa™ vaccines were administered intramuscularly into the right antero-lateral thigh, while the Rotarix™ vaccine was given orally.
  Interventions: Biological: DTPa-HBV-IPV/Hib; Biological: DTPa-IPV/Hib vaccine

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib — 1 intramuscular injection (3rd study vaccine dose)
  Other Names: INFANRIX HEXA™
Biological: DTPa-IPV/Hib vaccine — 3 intramuscular injections (1st, 2nd and 4th vaccine dose)

SUMMARY:
To assess the safety and reactogenicity of the DTPa-HBV-IPV/Hib vaccine and DTPa-IPV/Hib vaccine. This DTPa-IPV/Hib vaccine given at 3 and 4 months of age is co-administered with GSK Biologicals' rotavirus vaccine or Placebo. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Single group study. Subjects in GSK Biologicals' rotavirus study (Rota-028) in Singapore will be enrolled in this study.

ELIGIBILITY:
Inclusion criteria

* Subjects must have been enrolled in the Rota-028 study.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 11 and 17 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Subjects should have received two doses of hepatitis B vaccine: at birth and at approximately one month of age.

Exclusion criteria

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of the vaccine and ending 30 days after.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 702 (Actual)
Dates: Start 2003-12-01; Primary Completion 2007-02-01 (Actual); Study Completion 2007-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lim FS, Phua KB, Lee BW, Quak SH, Teoh YL, Ramakrishnan G, Han HH, Van Der Meeren O, Jacquets JM, Bock HL. Safety and reactogenicity of DTPa-HBV-IPV/Hib and DTPa-IPV/I-Hib vaccines in a post-marketing surveillance setting. Southeast Asian J Trop Med Public Health. 2011 Jan;42(1):138-47. PMID 21323176
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix Hexa Group: Healthy male or female subjects between and including 11 to 17 weeks of age, who were previously vaccinated with Rotarix in study 444563/028, additionally received 2 doses of Infanrix-IPV/Hib vaccine (at 3 and 4 months of age), 2 doses of Rotarix vaccine (at 2 and 4 months of age) and one dose of Infanrix Hexa vaccine (at 5 months of age) as a primary vaccination course, followed by administration of a booster dose of Infanrix-IPV/Hib vaccine (at 18 months of age). The Infanrix-IPV/Hib and Infanrix Hexa vaccines were administered intramuscularly into the right antero-lateral thigh, while the Rotarix vaccine was given orally.
Period: Overall Study
Arm/Group | Infanrix Hexa Group
Started | 702
Completed | 676
Not Completed | 26
Not completed — Lost to follow-up(complete vacc. course) | 13
Not completed — Migrated/moved from study area | 1
Not completed — Lost to follow-up(incompl. vacc. course) | 4
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 702
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 13.5 (0.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349
  Male | 353
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 1
  Japanese | 1
  Not specified | 27
  Chinese | 366
  Malay | 269
  Indian | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Assessed solicited local and general symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available and who filled in their symptom sheet.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 697
Participants
  Any Pain, Dose 1 | 130
  Any Redness, Dose 1 | 120
  Any Swelling, Dose 1 | 89
  Any Pain, Dose 2: number analyzed (Participants) | 695
  Any Pain, Dose 2 | 134
  Any Redness, Dose 2: number analyzed (Participants) | 695
  Any Redness, Dose 2 | 137
  Any Swelling, Dose 2: number analyzed (Participants) | 695
  Any Swelling, Dose 2 | 100
  Any Pain, Dose 3: number analyzed (Participants) | 661
  Any Pain, Dose 3 | 97
  Any Redness, Dose 3: number analyzed (Participants) | 661
  Any Redness, Dose 3 | 126
  Any Swelling, Dose 3: number analyzed (Participants) | 661
  Any Swelling, Dose 3 | 100
  Any Pain, Booster dose: number analyzed (Participants) | 565
  Any Pain, Booster dose | 166
  Any Redness, Booster dose: number analyzed (Participants) | 565
  Any Redness, Booster dose | 148
  Any Swelling, Booster dose: number analyzed (Participants) | 565
  Any Swelling, Booster dose | 115
  Any Pain, Across doses | 301
  Any Redness, Across doses | 273
  Any Swelling, Across doses | 215

2. Primary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 697
Participants
  Any Drowsiness, Dose 1 | 165
  Any Temperature (Axillary) (°C), Dose 1 | 139
  Any Irritability, Dose 1 | 229
  Any Loss of appetite, Dose 1 | 173
  Any Drowsiness, Dose 2: number analyzed (Participants) | 695
  Any Drowsiness, Dose 2 | 140
  Any Temperature (Axillary) (°C), Dose 2: number analyzed (Participants) | 695
  Any Temperature (Axillary) (°C), Dose 2 | 124
  Any Irritability, Dose 2: number analyzed (Participants) | 695
  Any Irritability, Dose 2 | 192
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 695
  Any Loss of appetite, Dose 2 | 155
  Any Drowsiness, Dose 3: number analyzed (Participants) | 661
  Any Drowsiness, Dose 3 | 106
  Any Temperature (Axillary) (°C), Dose 3: number analyzed (Participants) | 661
  Any Temperature (Axillary) (°C), Dose 3 | 100
  Any Irritability, Dose 3: number analyzed (Participants) | 661
  Any Irritability, Dose 3 | 161
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 661
  Any Loss of appetite, Dose 3 | 106
  Any Drowsiness, Booster dose: number analyzed (Participants) | 565
  Any Drowsiness, Booster dose | 89
  Any Temperature (Axillary) (°C), Booster dose: number analyzed (Participants) | 565
  Any Temperature (Axillary) (°C), Booster dose | 152
  Any Irritability, Booster dose: number analyzed (Participants) | 565
  Any Irritability, Booster dose | 163
  Any Loss of appetite, Booster dose: number analyzed (Participants) | 565
  Any Loss of appetite, Booster dose | 118
  Any Drowsiness, Across doses | 290
  Any Temperature (Axillary) (°C), Across doses | 330
  Any Irritability, Across doses | 381
  Any Loss of appetite, Across doses | 324

3. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 702
Participants | 321

4. Secondary Outcome: Number of Subjects Reporting Any Large Swelling Reactions
Description: A large swelling reaction was defined as swelling with a diameter greater than (>) 50 millimeters (mm), noticeable diffuse swelling or noticeable increase of limb circumference.
Time Frame: At Month 15, post-booster dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 702
Participants | 0

5. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 up to Month 21)
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 702
Participants | 108

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day (Days 0-3) post-vaccination period; Unsolicited AE(s): during the 30-day (Days 0-29) post-vaccination period; SAE(s): during the entire study period (Month 0 to Month 21).
Description: The occurrence of reported AEs (all/related) was not available and is encoded as equal to the number of subjects affected.
Arm/Group | Infanrix Hexa Group
All-Cause Mortality (participants affected / at risk) | 0/702
Serious Adverse Events (participants affected / at risk) | 108/702
Other Adverse Events (participants affected / at risk) | 594/702
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Hexa Group (N=702)
Head injury (Injury, poisoning and procedural complications) | 5
Foreign body trauma (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Febrile convulsion (Nervous system disorders) | 13
Convulsion (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Pyrexia (General disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1
Stag horn calculus (Renal and urinary disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Bronchiolitis (Infections and infestations) | 30
Gastroenteritis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 11
Gastritis viral (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Escherichia urinary tract infection (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 4
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 3
Hand-foot-and-mouth disease (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Abscess (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 2
Kawasaki's disease (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Abscess neck (Infections and infestations) | 1
Exanthema subitum (Infections and infestations) | 1
Herpangina (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Viral skin infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infanrix Hexa Group (N=702)
Pain (General disorders) | 301/697 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 273/697 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 215/697 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 290/697 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Fever (Axillary) (°C) (General disorders) | 330/697 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (General disorders) | 381/697 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 324/697 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Pyrexia (General disorders) | 46
Diarrhoea (Gastrointestinal disorders) | 40
Rash (Skin and subcutaneous tissue disorders) | 40
Upper respiratory tract infection (Infections and infestations) | 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.